CLINICAL TRIAL: NCT03571919
Title: Efficacy of Intravenous Lidocaine Infusion for Traumatic Rib Fracture Pain Control
Brief Title: Lidocaine Infusions for Rib Fractures
Acronym: Lidocare
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit during the Covid pandemic
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 44300
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Rib Fracture Multiple; Trauma Chest; Pain, Acute
Keywords: Lidocaine infusion
MeSH Terms: conditions — Thoracic Injuries; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Immediate care providers (nurses, primary teams) will be blinded; however, lidocaine levels will be monitored by the acute pain service, a consulting team providing direct care to the patient, who will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Will receive normal saline bolus and infusion and have sham lab draws every 8 hours.
  Interventions: Drug: Saline infusion
- Lidocaine (Active Comparator): Will receive lidocaine bolus and infusion and have lidocaine lab draws every 8 hours.
  Interventions: Drug: Lidocaine infusion

INTERVENTIONS:
Drug: Lidocaine infusion — Intravenous bolus of lidocaine (1.25 mg/kg) and then infusion at 1 mg/kg/hr
  Arms: Lidocaine
Drug: Saline infusion — Intravenous bolus of saline and then infusion
  Arms: Control

SUMMARY:
Patients with traumatic rib fractures not receiving regional anesthesia through a epidural or nerve block catheter will be recruited for the study. Once enrolled, they will be randomized to receive either intravenous lidocaine or intravenous saline for control of pain related to their rib fractures. In addition, they will receive other pain medications, such as acetaminophen, gabapentin, and opioid pain medications. Our primary outcome is a decrease in their opioid medication requirements.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 or older with 2+ rib fractures or > 65 with 2+ rib fractures Enrollment within 16 hours of admission Inability to receive epidural placement or other catheter-based regional anesthesia (coagulopathy, anticoagulation, bacteremia or infection over epidural site, patient refusal, vertebral fracture, spinal cord injury, inability to cooperate with procedure, BMI > 40) Isolated rib fracture (no other major injury or anticipation for invasive procedure)

Exclusion Criteria:

Inability to participate in traditional pain measures Severe alcohol withdrawal Chronic pain requiring opiates prior to admission GCS < 13 or inability to report pain Medical instability Positive pressure ventilation, either via non-invasive mask or endotracheal tube Hemodynamic instability or shock Flail chest with clinical evidence of paradoxical rib motion Contraindication to lidocaine History of or current bradycardia (HR < 50) or heart block (Mobitz II or 3rd degree) New onset or uncontrolled seizures Allergy to amide-type local anesthetic

Enrollment in other study that may affect the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Opioid pain medicine usage | Average per 24 hours
  Total opioid pain medicine usage

SECONDARY OUTCOMES:
PCA requirements | 5 days
  Percentage of patients requiring PCA
Pain score | 5 days
  Average pain scores
Length of stay | 5 days
  Average length of stay in ICU and hospital
Respiratory failure | 5 days
  Rates of pneumonia or other respiratory failure (pneumonia defined as (1) new pulmonary infiltrate on chest X-ray and (2) two of three of the following: (a) productive cough (b) WBC > 12,000 and (c) temperature > 38.0)
Death | up to 30 days
  Mortality rate between two groups
Mobility | 2 days
  Highest level of mobility on hospital day #2

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Choi, MD, Principal Investigator — Stanford University; Michael Y Lin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No